CLINICAL TRIAL: NCT00378976
Title: A Randomized, Double-blind, Placebo-controlled Crossover Trial of Valacyclovir for Suppression of HSV and HIV Shedding in HIV-1, HSV-2 Coinfected Men Who Have Sex With Men (MSM).
Brief Title: HSV-2 Suppression to Reduce HIV-1 Levels in HIV-1, HSV-2 Co-infected Men.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: GlaxoSmithKline (Industry); Asociación Civil Impacta Salud y Educación, Peru (Other)
Responsible Party: Connie Celum, MD, MPH, University of Washington
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 21760-A; AI277S7;AI38858;AI30731
Record Dates: First submitted 2006-09-19; First posted 2006-09-21 (Estimated); Last update posted 2013-08-22 (Estimated); Status verified 2013-08

CONDITIONS: HIV Infection; Herpes Simplex; Sexually Transmitted Diseases
Keywords: HIV infection; HIV shedding; HSV suppression; Co-infected; MSM; Reactivation; Valacyclovir
MeSH Terms: conditions — HIV Infections; Herpes Simplex; Sexually Transmitted Diseases | interventions — Valacyclovir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: valacyclovir
- 2 (Placebo Comparator)
  Interventions: Drug: matching placebo

INTERVENTIONS:
Drug: valacyclovir — 500 mg twice-daily oral
  Arms: 1
Drug: matching placebo — twice daily as per experimental drug
  Arms: 2

SUMMARY:
Over 80% of HIV-1 infected persons are also seropositive for HSV-2. Increasingly, clinical and epidemiologic evidence show the role of HSV in increasing HIV infectiousness. The evidence suggests that that HSV is an important cofactor in HIV transmission.

The trial's purpose is to assess the reduction in HIV shedding associated with valacyclovir for suppression of HSV-2 reactivation.

This proof-of-concept, randomized, double-blind, placebo controlled crossover trial of 20 HIV/HSV-2 co-infected men, assessed the effects of daily valacyclovir on HIV-1 levels in the plasma and rectal mucosa secretions.

DETAILED DESCRIPTION:
Herpes simplex virus type 2 (HSV-2) is common among HIV infected persons. HSV-2 reactivation is associated with increased plasma and genital HIV-1 levels, and in vitro, HSV-2 upregulates HIV transcription.

The trial assessed whether HSV-2 suppression reduces rectal and plasma HIV-1 levels in HIV-1, HSV-2 co-infected men who have sex with men (MSM).

Conducted in Lima Peru, 20 antiretroviral naive HIV-1 and HSV-2 seropositive MSM with CD4 >200 were randomly assigned to receive valacyclovir 500 mg bid or placebo for 8 weeks, than a 2 week washout period, followed by the alternative regimen for 8 weeks. Men collected daily home anogenital swabs for HSV DNA PCR, had three weekly anoscopy procedures for collection of rectal mucosal secretions for HIV-1 RNA, HSV DNA, and weekly plasma HIV-1 RNA by PCR. Outcomes were plasma and rectal HIV-1 levels by study arm.

ELIGIBILITY:
Inclusion Criteria:

* Greater than 18 years old,
* Documented HIV-1 seropositive,
* CD4 count greater than 200,
* Not on HIV antiretroviral therapy,
* HSV-2 seropositive as determined by Focus EIA (IN >3.5)
* Not intending to move out of the area for the duration of study participation.
* Willing and able to:provide independent written informed consent;undergo clinical evaluations;take study drug as directed;adhere to follow-up schedule.
* Bacterial STDs (symptomatic STD syndromes or laboratory-confirmed asymptomatic gonorrhea and syphilis) are treated within two weeks of study enrollment and random assignment.

Exclusion Criteria:

MSM who meet any of the following criteria are not eligible for this study:

* Known history of adverse reaction to valacyclovir, acyclovir or famciclovir;
* Planned open label use of acyclovir, valacyclovir, or famciclovir
* Known medical history of seizures
* Known renal failure, serum creatinine >2.0mg/dl
* Hematocrit < 30 %

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2003-08; Study Completion 2004-07 (Actual)

PRIMARY OUTCOMES:
Reduction in anogenital HIV-1 shedding with suppression of HSV-2 reactivation. | 18 weeks

SECONDARY OUTCOMES:
Evaluate HSV-2 suppression with decreased plasma HIV RNA levels | 18 weeks
Assess the effect of daily valacyclovir on pharyngeal shedding in HSV-1 seropositive individuals | 18 weeks
Determine the temporal pattern of HIV shedding in the rectum, pharynx and semen with respect to mucosal HSV-1 and HSV-2 reactivation; Determine HSV-2 suppression and HIV replication within rectal mucosa. | 18 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Connie Celum, MD, MPH, Principal Investigator — University of Washington
Locations (1):
- Asociacion Civil Impacta Salud y Educacion, Lima, Peru

REFERENCES:
- [Derived] Zuckerman RA, Lucchetti A, Whittington WL, Sanchez J, Coombs RW, Magaret A, Wald A, Corey L, Celum C. HSV suppression reduces seminal HIV-1 levels in HIV-1/HSV-2 co-infected men who have sex with men. AIDS. 2009 Feb 20;23(4):479-83. doi: 10.1097/QAD.0b013e328326ca62. PMID 19169140
- [Derived] Zuckerman RA, Lucchetti A, Whittington WL, Sanchez J, Coombs RW, Zuniga R, Magaret AS, Wald A, Corey L, Celum C. Herpes simplex virus (HSV) suppression with valacyclovir reduces rectal and blood plasma HIV-1 levels in HIV-1/HSV-2-seropositive men: a randomized, double-blind, placebo-controlled crossover trial. J Infect Dis. 2007 Nov 15;196(10):1500-8. doi: 10.1086/522523. Epub 2007 Oct 31. PMID 18008230